CLINICAL TRIAL: NCT02146274
Title: Observational Study of Patient-centered Research Into Outcomes Stroke Patients Prefer and Effectiveness Research
Brief Title: Patient-centered Research Into Outcomes Stroke Patients Prefer and Effectiveness Research
Acronym: PROSPER
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00049705
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Stroke; Ischemic Stroke
Keywords: PROSPER; Stroke; Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ischemic Stroke Patients: Patients who have had an ischemic stroke that are hospitalized in an acute-care setting.

SUMMARY:
PROSPER (Patient-centered Research into Outcomes Stroke patients Prefer and Effectiveness Research) is a three year research project to create a national, sustainable model to improve decision-making and patient-centered stroke outcomes through comparative effectiveness research.

DETAILED DESCRIPTION:
We propose to address existing evidence gaps and develop the requested data on the range of clinical outcomes that may be experienced by stroke survivors. To achieve these goals, we will link the nation's largest stroke registry, the American Heart Association (AHA) Get With The Guidelines-Stroke program and nationwide Medicare claims data, coupled with telephone interviews for longitudinal treatment and downstream patient-reported outcomes.

Design & Procedures:

Retrospective: Using GWTG-Stroke database and its associated 1900 hospitals, we will conduct several comparative research protocols prioritized by stroke survivor focus groups and surveys. GWTG-Stroke registry clinical data linked with Medicare claims will be used for analysis of effectiveness and safety of post-stroke therapies on long-term clinical outcomes (n= 450,000). Outcomes of interest include:

"Home-time" (days alive and at home) Death Stroke/TIA readmission All-cause readmission Cardiovascular readmission Bleeding readmission

Prospective:

We will use the existing AVAIL registry combined with an additional 2000 stroke survivors for a combined cohort of over 5000 patients to obtain detailed information on patient-reported outcomes. The AVAIL Registry (IRB # Pro00012243) collected data from 3000 stroke survivors between 2006 and 2008. We plan to use these data to supplement our prospective PROSPER study. The PROSPER study will enroll a minimum of 2,000 subjects to augment the data collected from the AVAIL study. Consented patients from at least 75 sites will complete interviews at 3 and 6 months after discharge. We anticipate that the PROSPER questionnaire will include the following tools: Fatigue Severity Scale (FSS), Patient Health Questionnaire (PHQ8), modified Rankin scale (mRS), Barthel Index, EuroQOL (EQ-5D), Stroke-specific quality of life (SSQOL-12) and Lawton Instrumental Activities of Daily Living (IADL). Sites will consent interested patients and have them complete a patient contact information form which includes, name, address, phone numbers, email address, etc. Outcomes of interest include: : Post-stroke fatigue, Depression, Chronic pain, Medication intolerance, Modified Rankin scale (mRS), EuroQOL and Stroke-specific quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Consistent with GWTG inclusion criteria, patients must be older than 18 and have a primary diagnosis of acute ischemic stroke.
* Ability to give informed consent or the availability of a surrogate who can consent on the patient's behalf.

Exclusion Criteria:

* Patients with subarachnoid or intracerebral hemorrhage
* Patients with transient ischemic attack (TIA)
* Patients with expected survival less than 6 months/discharged to hospice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ischemic Stroke patients
Sampling Method: Probability Sample
Enrollment: 1877 (Actual)
Dates: Start 2013-11; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernandez, MD, Principal Investigator — DCRI
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

REFERENCES:
- [Derived] Xian Y, Wu J, O'Brien EC, Fonarow GC, Olson DM, Schwamm LH, Bhatt DL, Smith EE, Suter RE, Hannah D, Lindholm B, Maisch L, Greiner MA, Lytle BL, Pencina MJ, Peterson ED, Hernandez AF. Real world effectiveness of warfarin among ischemic stroke patients with atrial fibrillation: observational analysis from Patient-Centered Research into Outcomes Stroke Patients Prefer and Effectiveness Research (PROSPER) study. BMJ. 2015 Jul 31;351:h3786. doi: 10.1136/bmj.h3786. PMID 26232340
- [Derived] Xian Y, O'Brien EC, Fonarow GC, Olson DM, Schwamm LH, Hannah D, Lindholm B, Maisch L, Lytle BL, Greiner MA, Wu J, Peterson ED, Pencina MJ, Hernandez AF. Patient-Centered Research into Outcomes Stroke Patients Prefer and Effectiveness Research: Implementing the patient-driven research paradigm to aid decision making in stroke care. Am Heart J. 2015 Jul;170(1):36-45, 45.e1-11. doi: 10.1016/j.ahj.2015.04.008. Epub 2015 Apr 18. PMID 26093862

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Observational survey
Groups:
- Ischemic Stroke Patients: Patients who have had an ischemic stroke
Period: Overall Study
Arm/Group | Ischemic Stroke Patients
Started | 1877
Completed | 1804
Not Completed | 73
Not completed — Protocol Violation | 73

BASELINE CHARACTERISTICS:
Population: Exclusions (Total N, # of sites, %, # excluded):
  1. Interviewed PROSPER patients with registry data 1,804 63
  2. Active patient status 1,715 62 95.1 -89
  3. Medical history panel >75% complete 1,652 60 96.3 -63
  4. Ischemic stroke as primary diagnosis 1,622 60 98.2 -30
  5. Exclude expired/left AMA/disposition UTD/missing 1,617 60 99.7 -5
Arm/Group | Ischemic Stroke Patients
Number analyzed (Participants) | 1617
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [55 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 760
  Male | 857
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race: white | 1229
  race: black | 227
  race: hispanic | 65
  race: asian | 32
  race: other/utd | 64
Antidepressant at Discharge [Count of Participants; unit: Participants]
  Antidepressant - Yes | 185
  Antidepressant - No | 1432

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: Patient Health Questionnaire - 2 Item (PHQ-2) Higher score suggests more depression; range of 0-6. A score of two or higher suggests a diagnosis of major depression.
Time Frame: 6 months after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ischemic Stroke Patients By Anti-depressant =Yes: Patients on Antidepressant at Discharge
- Ischemic Stroke Patients By Anti-depressant =No: Patients not on Antidepressant at Discharge
Arm/Group | Ischemic Stroke Patients By Anti-depressant =Yes | Ischemic Stroke Patients By Anti-depressant =No
Number analyzed (Participants) | 185 | 1432
units on a scale | .7 (.22) | .79 (.21)

2. Secondary Outcome: Functional Status
Description: Euro-QOL ver. 5D-3L (EQ 5D-3L) EQ-5D-3L Five level version of the Euro-QOL. Index Value ranging from 0-1.0 Higher scores indicate better functioning
Time Frame: 6 months after enrollment
Population: Comparing functional status of ischemic stroke patients who are and are not taking an antidepressant 6 months post enrollment
Measure: Median (Inter-Quartile Range); unit: score on scale
Groups:
- Ischemic Stroke Patients on Antidepressant (n=222): Ischemic stroke patients taking an antidepressant
- Ischemic Stroke Patients Not Taking an Antidepressant (n=760): Ischemic stroke patients not taking an antipressant.
Arm/Group | Ischemic Stroke Patients on Antidepressant (n=222) | Ischemic Stroke Patients Not Taking an Antidepressant (n=760)
Number analyzed (Participants) | 222 | 760
score on scale | 0.77 [0.47 to 0.83] | 0.83 [0.71 to 1]

ADVERSE EVENTS:
Time Frame: Not collected; observational study
Description: Not collected; observational study
Arm/Group | Ischemic Stroke Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
6 month prospective observational study. Patients not randomized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-02-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT02146274/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT02146274/SAP_001.pdf